CLINICAL TRIAL: NCT00567775
Title: Comparison of Pharmacokinetic Profiles of Human Soluble Insulin With Insulin Inhalation Solution in Paediatric Type 1 Diabetes Mellitus
Brief Title: Comparison of Human Insulin to Insulin Inhalation Solution in Children With Type 1 Diabetes
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Novo Nordisk A/S (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: NN1998-1274
Record Dates: First submitted 2007-11-30; First posted 2007-12-05 (Estimated); Last update posted 2017-03-01 (Actual); Status verified 2017-02

CONDITIONS: Diabetes; Diabetes Mellitus, Type 1
MeSH Terms: conditions — Diabetes Mellitus; Diabetes Mellitus, Type 1 | interventions — Insulin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Drug: human insulin
  Other Names: Actrapid®; Novolin® R
Drug: inhaled human insulin

SUMMARY:
This trial is conducted in Europe. The aim of this trial is to compare the pharmacokinetic profile of two different methods of insulin administration in children with type 1 diabetes.

ELIGIBILITY:
Inclusion Criteria:

* Type 1 diabetes
* Treatment for at least 12 months
* HbA1c lesser or equal to 11.0%
* Body weight between 25 and 80 Kg
* Capable to use the device

Exclusion Criteria:

* Any diseases other than diabetes requiring prescriptive medication
* Known or suspected allergy to trial product or related products
* Active proliferative retinopathy as judged by the Investigator
* Recurrent severe hypoglycaemia as judged by the Investigator
* The receipt of any investigational drug within 4 weeks prior to this trial

Ages: 6 Years to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 27 (Actual)
Dates: Start 2002-10-21 (Actual); Primary Completion 2002-11-20 (Actual); Study Completion 2002-11-20 (Actual)

PRIMARY OUTCOMES:
Area under the serum insulin curve | from 0 to 5 hours post-dosing

SECONDARY OUTCOMES:
Maximum serum insulin concentration | in the interval from 0 to 5 hours post-dosing
Time to maximum serum insulin concentration | in the interval from 0 to 5 hours post-dosing

CONTACTS AND LOCATIONS:
Overall Officials: Global Clinical Registry (GCR, 1452), Study Director — Novo Nordisk A/S
Locations (1):
- Novo Nordisk Investigational Site, Glostrup Municipality, Denmark

REFERENCES:
- See also: Clinical Trials at Novo Nordisk — http://novonordisk-trials.com